CLINICAL TRIAL: NCT00741494
Title: Effectiveness of the Use of the PICSI Dish (Hyaluronan Microdot) in the Selection of Sperm for Intracytoplasmic Sperm Injection (ICSI) for Patients Having a Low Versus High Proportion of Hyaluronan Binding Sperm (HBA)
Brief Title: Effectiveness of the Use of the PICSI Dish (Hyaluronan Microdot) in the Selection of Sperm for Intracytoplasmic Sperm Injection (ICSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biocoat (Industry)
Responsible Party: Kathryn Worrilow, Biocoat, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008PICSI03
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Male Factor Infertility
Keywords: infertility; ICSI; hyaluronan binding; sperm; sperm selection; male factor; hyaluronan; sperm maturity; clinical pregnancy rates; hyaluronan binding assay; HBA; PICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (No Intervention): HBA score over 65% control
- 2 (No Intervention): HBA score over 65%, non-participant (to even out the participation between patients with low HBA scores and those with high HBA scores)
- 3 (Active Comparator): HBA score over 65%. PICSI dish is used to select the sperm for ICSI.
  Interventions: Device: PICSI dish
- 4 (Experimental): HBA score less than 65%. PICSI dish used to select sperm for ICSI.
  Interventions: Device: PICSI dish
- 5 (No Intervention): HBA Score less than 65%. Control

INTERVENTIONS:
Device: PICSI dish — Sperm are added to the PICSI dish. Only those that bind to the hyaluronan microdots are selected for ICSI
  Arms: 3; 4

SUMMARY:
The purpose of this study is to determine if using microdots of hyaluronan (PICSI) to select sperm for ICSI will result in increased pregnancies especially with men that have a low hyaluronan binding score (HBA).

ELIGIBILITY:
Inclusion Criteria:

* IVF patients who require the ICSI procedure and whose care is being managed by the clinical and scientific staff of the participating groups, will be included in the study.

Exclusion Criteria:

* IVF patients who do not require the ICSI procedure will be excluded from the study. In addition the following groups of patients will also be excluded:

  * Patients using testicular sperm.
  * Patients using donor sperm.
  * Patients where the female partner is over 40 years of age
  * Patients who have an initial HBA score less than or equal to 2%
  * Patients who have a sperm count less than or equal to 10,000 motile sperm per ml.
  * Patients who produce less than 4 Metaphase II oocytes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 801 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 8 weeks post ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Worrilow, Ph.D., Study Director — Biocoat
Locations (9):
- United States (9):
  - Huntington Reproductive Center, Laguna Hills, California
  - Reproductive Science Center of the Bay Area, San Ramon, California
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Reproductive Biology Associates, Atlanta, Georgia
  - Fertility Centers of Illinois, Chicago, Illinois
  - CNY Fertility Center, Syracuse, New York
  - Abington IVF and Genetics Toll Center for Reprodcution, Abington, Pennsylvania
  - Center for Reproduction and Infertility, Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Seattle Reproductive Medicine, Seattle, Washington

REFERENCES:
- [Derived] Worrilow KC, Eid S, Woodhouse D, Perloe M, Smith S, Witmyer J, Ivani K, Khoury C, Ball GD, Elliot T, Lieberman J. Use of hyaluronan in the selection of sperm for intracytoplasmic sperm injection (ICSI): significant improvement in clinical outcomes--multicenter, double-blinded and randomized controlled trial. Hum Reprod. 2013 Feb;28(2):306-14. doi: 10.1093/humrep/des417. Epub 2012 Nov 30. PMID 23203216